CLINICAL TRIAL: NCT06988436
Title: FETAL PULMONARY VEIN AND UMBILICAL ARTERY PULSATILITY INDICES AS PREDICTORS OF FETAL GROWTH RESTRICTION IN DIABETIC AND HYPERTENSIVE PREGNANT WOMEN
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Other Study IDs: 365
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertensive group: Pregnant women diagnosed with preexisting or gestational hypertension
  Interventions: Diagnostic Test: Ultrasound
- Diabetic group: Pregnant women diagnosed with preexisting or gestational diabetes
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — All the participants were scanned using B mode sonography to determine the fetal biometric parameters (BPD, HC, AC and FL). The machine automatically calculated the estimated fetal weight using the Headlock formula. umbilical artery pulsatility index (UAPI) and pulmonary vein pulsatility index (PVPI) were measured in the study

SUMMARY:
Diabetic and hypertensive pregnant women attending at Kasr Alani for antenatal care were subjected to Complete History taking. All the participants were scanned using B mode sonography to determine the fetal biometric parameters (BPD, HC, AC and FL).Only umbilical artery pulsatility index (UAPI) and pulmonary vein pulsatility index (PVPI) were measured in the study. UAPI and PVPI were measured between 28 and 34 weeks of gestation at the first routine ultrasound scheduled.

DETAILED DESCRIPTION:
Diabetic and hypertensive pregnant women attending at Kasr Alani for antenatal care were subjected to Complete History taking. All the participants were scanned using B mode sonography to determine the fetal biometric parameters (BPD, HC, AC and FL).Only umbilical artery pulsatility index (UAPI) and pulmonary vein pulsatility index (PVPI) were measured in the study. UAPI and PVPI were measured between 28 and 34 weeks of gestation at the first routine ultrasound scheduled. The umbilical artery Doppler examinations were conducted on a free-floating loop at the middle of the cord, away from its placenta and fetal abdominal insertion sites. The Doppler angle was <60°, for an optimal Doppler signal. The recording was done when fetal breathing movement or uterine contraction was absent. The Doppler wall filter was set at 50 - 100Hz, spectral peak average intensities were below 100 m/wcm2, and pulsed Doppler sample gate size was 2 mm (Adedo et al., 2022). The following umbilical artery Doppler indices (UADI) were calculated automatically by the machine: Peak Systolic Velocity (PSV) in cm/s, End Diastolic Velocity (EDV) in cm/s, Pulsatility Index (PI), Resistive Index (RI), and Systolic/Diastolic Ratio (S/D Ratio). The umbilical artery waveform pattern was also analyzed and classified into: normal diastolic flow, reduced diastolic flow, absent diastolic flow and reversed diastolic flow. The values of UAPI considered abnormal if >95th percentile are as follows: at 28th Wk. > 1.35, 29th Wk. >1.32, 30th Wk. >1.29, 31stWk >1.27, 32ndWk. >1.25, 33thWk >1.22 and 34th Wk >1.2 (Adedo et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18 and 44 years.
* Gestational age: 28 - 34 weeks of gestation at time of examination (only women with confirmed GA by sure LMP and/or first trimester US scan).
* Singleton pregnancy.
* Hypertensive women (preexisting or gestational hypertension).
* Diabetic women (preexisting or gestational diabetes).

Exclusion Criteria:

* Women with any medical disorder (apart from diabetes and hypertension).
* Women with multiple pregnancies.
* Women with inadequate ultrasound images (i.e., marked obesity).
* Women with fetuses with chromosomal abnormalities or congenital anomalies and other factors that could affect fetal growth.
* Unavailable perinatal outcome data

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Diabetic and hypertensive pregnant women attending at Kasr Alani for antenatal care with the following criteria.
  Women were divided into 2 equal groups (total 82 cases):
  * Group A: hypertensive group 41 patients.
  * Group B: diabetic group 41 patients.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Prediction of fetal growth restriction | At time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided